CLINICAL TRIAL: NCT04734327
Title: Orthokine Therapy in Lumbar Degenerative Disease: Does the Route of Administration Really Matter
Brief Title: Orthokine Therapy in Lumbar Degenerative Disease
Acronym: OLDDD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sutherland Medical Center (Other)
Responsible Party: Principal Investigator, Piotr Godek, Principal Investigator, Sutherland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC2021001
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Degenerative Disc Disease; Lumbar Region
Keywords: degenerative disc disease; lumbar spine; conservative treatment; Orthokine
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthokine periradicular injection (Experimental): Ultrasound guided injections
  Interventions: Procedure: Orthokine periradicular injection
- Orthokine epidural injection (Active Comparator): Ultrasound guided injections
  Interventions: Procedure: Orthokine epidural injection

INTERVENTIONS:
Procedure: Orthokine periradicular injection — Ultrasound guided injections
  Arms: Orthokine periradicular injection
Procedure: Orthokine epidural injection — Ultrasound guided injections
  Arms: Orthokine epidural injection

SUMMARY:
The aim of the trial is the comparison of the effectiveness of two methods of Orthokine administration (periradicular or epidural) in lumbar degenerative disc disease.

DETAILED DESCRIPTION:
BACKGROUND: Lumbar Degenerative Disc Disease (LDDD) is a serious, global health problem for patients from the third decade of life. It is assumed that 75-85% of the population suffer from pain in the lumbar spine at least once during their lifetime (vital morbidity), and 3-5% of the population suffer from root-type pain.

The annual prevalence of the spine complaints in the United States alone ranges from 15 to 20%, and in Europe it ranges from 25 to 45%.

In addition to the immeasurable losses associated with impaired patient activity and a significant reduction in the quality of their life, LBP is the greatest burden for the world economy, measured by the years lived with disability (YLD) index due to a significant reduction in the productivity and professional ability of patients affected by LBP.

AIM: Assessment of the effectiveness of symptomatic treatment of Lumbar Degenerative Disc Disease (LDDD) with the autologous Orthokine serum, comparison of two methods of its application - epidural or periradicular.

DESIGN: Randomized prospective trial without blinding SETTING: Open study for outpatients, single center study POPULATION: local population METHODS: Two groups of patients (A, B) with confirmed LDDD by MRI, without gender or age limitation, meeting the health conditions according to the inclusion and exclusion criteria. There will be 50 people in each group (100 people in total).

Group A - therapy with Orthokine serum - a total of 4 injections of 2 doses at weekly intervals (4 doses of 4 ml of serum in total), injections will be performed into the epidural space from an interlaminar access under ultrasound guidance by the same operator.

Group B - therapy with Orthokine serum - a total of 4 injections of 1 or 2 doses depending on the number of levels occupied at weekly intervals (a total of 4 doses of 4 ml of serum), injections will be performed periradicular (transforaminal) under ultrasound guidance by the same operator.

Assessment tools: Numeric Rating Scale NRS (0-10), Oswestry Disability Index questionnaire, Roland Morris questionnaire, EQ-5D-5L questionnaire Control points W0 - before the therapy, W1 - 1 month after the last dose of serum W2 - 3 months after the last dose of serum W3 - 6 months after the last serum dose.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical symptoms of LDDD in the lumbar region
2. LDDD confirmed by MRI
3. No contraindications to injections (hemorrhagic diathesis, anticoagulants, skin lesions)
4. An adult consenting to participate in the study

Exclusion Criteria:

1. Presence of severe neurological deficits requiring surgery
2. Discopathy of other origin - traumatic, spondylolisthesis, cancer, infection, inflammatory systemic diseases
3. Previous surgical treatment in the lumbar spine
4. Mental state that prevents cooperation during injection
5. Contraindications for injection (hemorrhagic diathesis, anticoagulants, skin lesions)

5. Lack of consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in EQ-5D-5L index from baseline to 24 weeks | Time Frame: Change from baseline to 24 weeks
  EQ-5D-5L index estimated from EQ-5D-5L descriptive system based on Polish directly measured value set. Minimum: -0.590; Maximum: 1.0; More points means better outcome.
Change in Oswestry Disability Index from baseline to 24 weeks | Time Frame: Change from baseline to 24 weeks
  Disease-specific questionnaire. Range: 0 (the best score) - 50 (the worst score).
Change in Roland Morris Questionnaire score from baseline to 24 weeks | Time Frame: Change from baseline to 24 weeks
  Disease-specific questionnaire. Range: 0 (the best score) - 24 (the worst score).

SECONDARY OUTCOMES:
Pain according to Numeric Rating Scale (NRS) from baseline to 4 weeks | Change from baseline to 4 weeks
  0 (no pain) - 10 points (the worst possible pain)
Pain according to Numeric Rating Scale (NRS) from baseline to 12 weeks | Change from baseline to 12 weeks
  0 (no pain) - 10 points (the worst possible pain)
Pain according to Numeric Rating Scale (NRS) from baseline to 24 weeks | Change from baseline to 24 weeks
  0 (no pain) - 10 points (the worst possible pain)
Change in EQ-5D-5L index from baseline to 4 week | Change from baseline to 4 weeks
  EQ-5D-5L index estimated from EQ-5D-5L descriptive system based on Polish directly measured value set. Minimum: -0.590; Maximum: 1.0; More points means better outcome.
Change in EQ-5D-5L index from baseline to 12 week | Change from baseline to 12 weeks
  EQ-5D-5L index estimated from EQ-5D-5L descriptive system based on Polish directly measured value set. Minimum: -0.590; Maximum: 1.0; More points means better outcome.
Change in Oswestry Disability Index from baseline to 4 weeks | Change from baseline to 4 weeks
  Disease-specific questionnaire. Range: 0 (the best score) - 50 (the worst score).
Change in Oswestry Disability Index from baseline to 12 weeks | Change from baseline to 12 weeks
  Disease-specific questionnaire. Range: 0 (the best score) - 50 (the worst score).
Change in Roland Morris Questionnaire score from baseline to 4 weeks | Change from baseline to 4 weeks
  Disease-specific questionnaire. Range: 0 (the best score) - 24 (the worst score).
Change in Roland Morris Questionnaire score from baseline to 12 weeks | Change from baseline to 12 weeks
  Disease-specific questionnaire. Range: 0 (the best score) - 24 (the worst score).

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Godek, PhD, Principal Investigator — Sutherland Medical Center
Locations (1):
- Sutherland Medical Center, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No